CLINICAL TRIAL: NCT05885581
Title: Grow Well/Crecer Bien: Addressing Childhood Obesity in Low-income Families
Brief Title: "Grow Well: Addressing Childhood Obesity in Low-income Families"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Riverside (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: UCRiverside
Record Dates: First submitted 2023-04-13; First posted 2023-06-02 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Diet Habit
MeSH Terms: conditions — Feeding Behavior | interventions — Methods; Control Groups

STUDY DESIGN:
Intervention Model Description: The goal of the research is to provide nutrition education on healthy infant feeding to reduce risk for early childhood obesity. The prevalence of obesity in early life remains unacceptably high, especially among low-income children, most are ethnic minorities. Marked ethnic disparities are evident by two years of age, which suggests that existing interventions are not adequate. Early prevention is critical, especially for low-income children.
  This project, which focuses on an-at-risk child population, has great potential to address our nation's growing crisis of childhood obesity, which can dramatically improve the health of millions of low-income children, their families, and their future children.
Who Masked: Care Provider
Masking Description: Randomization will occur once base-line data is collected. Comparisons will be made between the intervention and control groups during the first 6 months of the intervention. The focus is on Latinx Spanish-speaking families; however, all our material is in English and Spanish to accommodate language preferences. Additionally, if a mother or caregiver prefers Purépecha, a language commonly spoken in the region, a Purépecha-speaking team member can translate orally from Spanish to Purépecha as this is an oral and not written language.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Grow Well and will receive the adapted Healthy Beginnings Curriculum (n= 15 mother-infant-caregiver triad) determine the feasibility, acceptability, and preliminary efficacy of the adapted intervention. The intervention will be on mothers' and caregivers' infant feeding knowledge, use of recommended feeding practices, and infant anthropometric measurement outcomes.
  Interventions: Other: Arm A Grow Well
- Group B: (Active Comparator): Group B will receive the Healthy Steps curriculum or treatment as usual as this is the curriculum commonly shared during well baby visits (n= 15 mother-infant-caregiver triad).
  Interventions: Other: Arm B Healthy Steps

INTERVENTIONS:
Other: Arm A Grow Well — 1. the preliminary efficacy of the adapted intervention on mothers' and caregivers' infant feeding knowledge, use of recommended feeding practices, and infant anthropometric measurement outcomes.
  2. the feasibility of implementing the intervention and its acceptability among mothers and caregivers.
  3. the feasibility of collecting infant anthropometric data.
  Other Names: Intervention
  Arms: Group A
Other: Arm B Healthy Steps — Group B: Healthy Steps and will receive the Healthy Steps curriculum or treatment as usual as this is the curriculum commonly shared during well baby visits (n= 15 mother-infant-caregiver triad).
  Other Names: Control Group
  Arms: Group B:

SUMMARY:
This research uses community based participatory research (CBPR) to engage low-income Latinx families in research to pilot test an adapted nutrition education program compared to an existing nutrition education program. The goal of the research is to provide nutrition education on healthy infant feeding to reduce risk for early childhood obesity. The prevalence of obesity in early life remains unacceptably high, especially among low-income children, most are ethnic minorities. Marked ethnic disparities are evident by two years of age, which suggests that existing interventions are not adequate. This project, which focuses on an-at-risk child population, has great potential to address our nation's growing crisis of childhood obesity, which can dramatically improve the health of millions of low-income children, their families, and their future children.

DETAILED DESCRIPTION:
This research will implement and evaluate an existing healthy infant feeding intervention, Healthy Beginnings, which was developed for English-speaking low-income mothers in Australia and delivered by public health nurses via in-home visits. The investigator will test the efficacy of an adapted version of this intervention in comparison to the original intervention.

Aim 1. Pilot test an adapted nutrition education program of, compared to the original program curriculum.

● Using a pilot randomized control trial with 30 mother-infant-caregiver triad (15 intervention, 15 control) determine the feasibility, acceptability, and preliminary efficacy of the adapted intervention compared to the original intervention.

The investigator hypothesize that the adapted intervention will be feasible, acceptable to study participants, and efficacious in addressing feeding styles and practices and caregivers' role in infant feeding. The investigator anticipate that the intervention will be feasible to deliver and acceptable to mothers' participants and caregivers' participants, and that the mother's participants-infant-caregiver triads randomized to intervention with the adapted Healthy Beginnings curriculum compared to the treatment as usual control group will demonstrate greater improvements in outcomes (i.e., infant feeding knowledge and use of recommended feeding practices) after 6 months compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Identify as Latina Mothers with infant who identified as caregivers.
* 18 years or older.
* Speak English, Spanish or Purépecha.
* Mother (biological, adoptive, foster) of an infant ages 4 months or younger, who had a normal birth weight (greater than or equal to 5. lbs., 8 oz.)
* Live in Inland Southern California.
* Income eligible (mothers or their children) for government programs such as WIC, Early Head Start, MediCal, CalFresh and similar programs.
* Willing to have a community health worker enter your home to provide 30-45 minute in person sessions once per month over 6 months.
* Have another caregiver 18 years or older who participates in at least 3 hours of care per week and agrees to participate in the home sessions.

Exclusion Criteria:

* Individual not willing to sign informed consent.
* Unable to speak English, Spanish or Perepecha.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Females
Enrollment: 96 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Efficacy of the adapted intervention on mothers' and caregivers' infant. | 0 months (infant birth) to one year
  It will include an intervention and control group and will be carried out over 6 months or 24 weeks and will involve 30 mother-infant-caregiver triads. Pretest and posttest surveys will be collected at baseline (week 1), and at six months follow up (week 24).
Data Collection-Infant Feeding Practices | 0 months (infant birth) to one year
  The survey will collect data on infant feeding practices using the validated Infant Feeding Scale Questionnaire (Thompson et al., 2009). It questionnaire is designed to assess maternal attitude towards infant feeding methods and to predict breastfeeding intention and exclusivity. The scale is composed of 17 items with a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree).The measurements of unit will be in fluid ounces.
Data collection-anthropometric data | 0 months (infant birth) to one year
  The study team members will collect anthropometric data, weight, length, and body fat composition from infants at the beginning and end of the study period. The infant body fat composition using fat calipers; Skinfolds (mm) Triceps (mm); Subscapular (mm); Liver (mm); Flank(mm); Thigh (mm)
Data collection-anthropometric data | 0 months (infant birth) to one year
  The study team members will collect anthropometric data, weight, length, and body fat composition from infants at the beginning and end of the study period. The infant weight using Body measurements: Child Weight (kg)
Data collection-anthropometric data | 0 months (infant birth) to one year
  The study team members will collect anthropometric data, weight, length, and body fat composition from infants at the beginning and end of the study period. The infant length using an infant measuring device that infants lay on, and body fat composition using fat calipers. Length (cm).
Data collection-sociodemographic questions | 0 months (infant birth) to one year
  The study team members will collect data Socio-demographic variables include, for example, age, sex, education, migration background and ethnicity, religious affiliation, marital status, household, employment, and income.

CONTACTS AND LOCATIONS:
Locations (1):
- UC Riverside, Riverside, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-04-05): https://cdn.clinicaltrials.gov/large-docs/81/NCT05885581/Prot_000.pdf
  • Informed Consent Form (2023-04-05): https://cdn.clinicaltrials.gov/large-docs/81/NCT05885581/ICF_001.pdf